CLINICAL TRIAL: NCT03812822
Title: The Effects of Using Insoles on Walking in Children With Increased Femoral Anteversion and Pes Planovalgus
Brief Title: Describing the Effects of Insoles in Children With Increased Femoral Anteversion and Pes Planovalgus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Kültür University (Other)
Responsible Party: Principal Investigator, Halenur Evrendilek, Research Assistant, Istanbul Kültür University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018/376
Record Dates: First submitted 2019-01-17; First posted 2019-01-23 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2019-01

CONDITIONS: Femoral Anteversion; Pes Planovalgus; Flat Foot
Keywords: Femoral anteversion, flat foot, insole, gait
MeSH Terms: conditions — Clubfoot; Flatfoot | interventions — Foot Orthoses

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insole Group (Experimental): Gait and foot posture analysis with and without the insole.
  Interventions: Device: Insole
- Control Group (No Intervention): Gait and foot posture analysis.

INTERVENTIONS:
Device: Insole — Custom-made insoles which support the foot at subtalar neutral position
  Arms: Insole Group

SUMMARY:
Increased Femoral Anteversion is a transverse plan problem that affects lower body alignment, walking and standing characteristics and also pes planovalgus mostly accompanies with IFA. It is shown that children with IFA and PPV have back and leg pain, fatigue, muscle cramps and they are under the risk for chronic disorders such as osteoarthritis, scoliosis and muscle injuries.

Insoles, which reduce pronation of foot (flat foot), provide apparently a static correction by supporting proper alignment in children with IFA and PPV. However, the dynamic effects of insoles to lower extremity biomechanics while walking is not known.

The aims of this study are to determine the effects of the insoles on walking biomechanics in children with IFA and PPV by comparing with their healthy peers.

ELIGIBILITY:
Inclusion Criteria:

* Insole Group Between the ages 7-15, Trochanteric Prominens Angle Test > 20⁰, Hip internal rotation angle > 60⁰, Without insole Foot Posture Index score > 5, With insole Foot Posture Index score > 4, Using their insoles' at least one month.
* Control Group Between the ages 7-15, Trochanteric Prominens Angle Test < 20⁰, Foot Posture Index score < 5, Without any neurologic or orthopedic disease

Exclusion Criteria:

Neurological and / or musculoskeletal problems, Orthopedic problems to prevent walking.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-24 (Actual); Study Completion 2019-12-24 (Actual)

PRIMARY OUTCOMES:
Gait Analysis | Day 1
  Three-dimensional gait analysis (Temporo-spatial parameters and pelvis, hip, knee and ankle kinematic in three plans)
Static Foot Posture Assesment | Day 1
  Foot Posture Index - 6 6 items ( 1.talar head palpation, 2.supra and infra lateral malleolar curvature,3.calcaneal frontal plane position, 4.prominence in the region of the talonavicular joint, 5.congruence of the medial longitudinal arch, and 6.abduction/adduction of the forefoot on the rearfoot)

CONTACTS AND LOCATIONS:
Overall Officials: Halenur Evrendilek, GRAD ASST, Study Chair — İstanbul Kültür University; Ekin Akalan, PROF, Study Director — İstanbul Kültür University; Miray Budak, ASST PROF, Study Director — İstanbul Medipol University
Locations (2):
- Turkey (Türkiye) (2):
  - İstanbul Kültür Üniversitesi, Istanbul
  - İstanbul University, Faculty of Medicine, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided